CLINICAL TRIAL: NCT02114216
Title: Symptomatic Gastroesophageal Reflux Disease is Associated With Increased TRPV1 and PAR2 mRNA Expression Levels in the Esophageal Mucosa
Brief Title: Nociceptors, Neurotrophic Factors and Cytokine Expression in Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B-1211/180-003
Record Dates: First submitted 2014-03-23; First posted 2014-04-15 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Gastro-esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (Sham Comparator): Subjects who do not show mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and do not complain of GERD symptoms. Endoscopic mucosal biopsy was done for every subject.
  Interventions: Procedure: endoscopic mucosal biopsy
- ERD group (Active Comparator): Subjects who have mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and/or complain of GERD symptoms. Endoscopic mucosal biopsy was done for every subject.
  Interventions: Procedure: endoscopic mucosal biopsy
- NERD group (Active Comparator): Subjects who do not have mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and complain of GERD symptoms. Endoscopic mucosal biopsy was done for every subject.
  Interventions: Procedure: endoscopic mucosal biopsy

INTERVENTIONS:
Procedure: endoscopic mucosal biopsy — endoscopic mucosal biopsy was undertaken for every participant.

SUMMARY:
Transient receptor potential vanilloid-1 (TRPV1) receptor and proteinase-activated receptor 2 (PAR2) have been implicated in the mechanism of acid induced inflammation in gastroesophageal reflux disease (GERD). We aimed to evaluate TRPV1 and PAR2 mRNA expression levels in the GERD patients and their relationship with endoscopic findings and reflux symptoms.

DETAILED DESCRIPTION:
All the subjects receive upper GI endoscopy and completed questionnaires about GERD symptoms under the supervision of a well-trained interviewer. Subjects are excluded if there was a history of gastrointestinal surgery, Barrett's esophagus, esophageal motility disorder, duodenal ulcer, benign gastric ulcer or gastroduodenal cancer and if he or she had any history of systemic disease requiring chronic medication (except for hypertension and diabetes mellitus).

The subjects are classified into 3 groups after upper GI endoscopy and completing questionnaires about GERDsymptoms ; ERD(erosive reflux disease), NERD(nonerosive reflux disease) and control group.

ELIGIBILITY:
Inclusion Criteria:

* subjects who completed upper GI endoscopy and questionnaires about GERD symptoms

Exclusion Criteria:

* a history of gastrointestinal surgery
* Barrett's esophagus
* esophageal motility disorder
* duodenal ulcer
* benign gastric ulcer
* gastroduodenal cancer
* if he or she had any history of systemic disease requiring chronic medication (except for hypertension and diabetes mellitus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Principal Investigator — Professor
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were enrolled prospectively at Seoul National University Bundang Hospital between March 2010 and August 2014. Those enrolled subjects visited SNUBH gastroenterology department mainly for evaluating the origin of suspicious GERD symptoms or for screening of gastric cancer.
Pre-assignment Details: Subjects were excluded if there was a history of gastrointestinal surgery, Barrett's esophagus, esophageal motility disorder, duodenal ulcer, benign gastric ulcer or gastroduodenal cancer and any history of systemic disease requiring chronic medication (except for hypertension and diabetes mellitus).
Groups:
- Control Group: subjects who do not show mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and do not complain of GERD symptoms
- ERD Group: subjects who have mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and/or complain of GERD symptoms
- NERD Group: subjects who do not have mucosal breaks in the upper GI endoscopy consistent with reflux esophagitis and complain of GERD symptoms
Period: Overall Study
Arm/Group | Control Group | ERD Group | NERD Group
Started | 16 | 45 | 14
Completed | 16 | 45 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | ERD Group | NERD Group | Total
Number analyzed (Participants) | 16 | 45 | 14 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.6) | 52.3 (10.39) | 52.7 (13.8) | 52.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 22 | 7 | 38
  Male | 7 | 23 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: TRPV1, GDNF, and NGF mRNA Expression of Esophageal Mucosa
Description: The primers used in real-time qPCR were designed using PrimerExpress Software V2.0 (Applied Biosystems, Foster City, CA, USA) based on sequence information from the National Center for Biotechnology Information database. Real-time qPCR was performed in triplicate by using a StepOnePlus Real-time PCR (Applied Biosystems) with SYBR Premix Ex TaqTM (Takara Bio, Shiga, Japan) according to manufacturers' instructions and protocols. Thermal cycling was performed as follows: initial denaturation at 95 °C for 10s followed by 40 cycles of 95 °C for 5 s and 60 °C for 33s. Homo b-actin was used as a reference; i.e. each sample was normalized on the basis of its b-actin content. The relative change in all target genes expression was determined by the fold-change analysis.
Time Frame: up to 24weeks
Measure: Mean (Standard Error); unit: Fold change
Arm/Group | Control Group | ERD Group | NERD Group
Number analyzed (Participants) | 16 | 45 | 14
Fold change
  TRPV1 | 1.14 (0.25) | 3.25 (0.32) | 2.33 (0.22)
  GDNF | 1.39 (0.35) | 2.47 (0.33) | 2.05 (0.16)
  NGF | 1.62 (0.37) | 2.65 (0.21) | 2.29 (0.13)

2. Secondary Outcome: PAR2 and IL-8 Expression of Esophageal Mucosa
Description: as for outcome 1
Time Frame: up to 24weeks
Measure: Mean (Standard Error); unit: Fold change
Arm/Group | Control Group | ERD Group | NERD Group
Number analyzed (Participants) | 16 | 45 | 14
Fold change
  PAR2 | 1.37 (0.20) | 2.42 (0.17) | 2.29 (0.36)
  IL8 | 2.01 (0.60) | 4.36 (0.32) | 4.01 (0.35)

ADVERSE EVENTS:
Description: Serious and/or other[non-serious] adeverse events were not collected/assessed.
Arm/Group | Control Group | ERD Group | NERD Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No